CLINICAL TRIAL: NCT05491915
Title: The MONARCH (Multicenter Occipital Neuralgia and Cervicogenic Headache) Case Series Study: Treatment of Head Pain With the SPRINT® Peripheral Nerve Stimulation (PNS) System
Brief Title: The MONARCH Case Series Study: SPRINT® Peripheral Nerve Stimulation for the Treatment of Head Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0156-CSP-000
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cervicogenic Headache; Occipital Neuralgia
Keywords: Electrical Stimulation; Neuromodulation; Head pain; Headache; Neck pain
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Neck Pain | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Peripheral Nerve Stimulation (Experimental): All study subjects will have up to 2 leads placed in the back of their neck, will use the SPRINT Peripheral Nerve Stimulation (PNS) System, and will receive electrical stimulation.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System delivers mild electrical stimulation to the occipital nerves. The SPRINT System includes up to two leads (small wires) that are placed through your skin at the top of your neck. The leads attach to devices worn on your body that deliver stimulation (called Stimulators).

SUMMARY:
The purpose of this study is to learn if pain can be relieved by delivering small amounts of electricity (called "electrical stimulation") to the nerves at the top of the neck. This study will use a device called the SPRINT® PNS System. PNS stands for peripheral nerve stimulation (PNS). This device is cleared by the FDA for up to 60 days of use for relief of chronic or acute pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed cervicogenic headache (CGH) or occipital neuralgia (ON)

Key Exclusion Criteria:

* Prior cervical or cranial occipital surgery
* Implanted electronic device (dependent on implant's intended treatment, location, and electrical current pathway)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in average pain and/or reduction in pain interference. | Up to 8-weeks after Start of Therapy (SOT)
  Average pain is measured using question 5 from the Brief Pain Inventory-Short Form (BPI-5) and pain interference is measured using question 9 from the Brief Pain Inventory-Short Form (BPI-9). BPI-5 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain. BPI-9 is a scale of 0 to 10 where 0 represents no interference and 10 represents complete interference.
Study-Related Adverse Events (AEs) | During the Lead Placement procedure (SOT)
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 24-48 hours post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 1-week post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 2-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 3-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 4-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 5-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 6-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 7-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 8-weeks post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 3-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 6-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 9-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 12-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 18-months post-SOT
  Occurrence and type of study-related AEs
Study-Related Adverse Events (AEs) | 24-months post-SOT
  Occurrence and type of study-related AEs

SECONDARY OUTCOMES:
Reduction in average pain intensity | Baseline, 8-weeks after SOT, 3-months after SOT, 6-months after SOT, 9-months after SOT, 12-months after SOT
  Average pain scores measured using question 5 from the Brief Pain Inventory- Short Form.
Reduction in pain interference | Baseline, 8-weeks after SOT, 3-months after SOT, 6-months after SOT, 9-months after SOT, 12-months after SOT
  Average pain interference scores measured using question 9 from the Brief Pain Inventory- Short Form.
Reduction in pain medication usage | Baseline, 8-weeks after SOT, 3-months after SOT, 6-months after SOT, 9-months after SOT, 12-months after SOT
  Analgesic medication consumption will be collected.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pacific Research Institute, Santa Rosa, California
  - MedVadis Research, Waltham, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Center of Clinical Research, Winston-Salem, North Carolina
  - Pain Specialists of America - South Austin - James Casey, Austin, Texas
  - Pain Specialists of America - Cedar Park, Cedar Park, Texas
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Pain Specialists of America - Round Rock, Round Rock, Texas
  - Pain Specialists of America - San Marcos, San Marcos, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Website — http://www.sprintpns.com